CLINICAL TRIAL: NCT01850823
Title: Clinical Equivalence Study of Mometasone Nasal Spray
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Collaborators: Watson Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71209805
Record Dates: First submitted 2013-05-06; First posted 2013-05-10 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- NASONEX® Nasal Spray (Schering Corporation) (Active Comparator): Mometasone Nasal spray
  Interventions: Drug: Mometasone Nasal Spray
- Mometasone Nasal Spray (Watson Laboratories, Inc) (Experimental): Mometasone Nasal spray
  Interventions: Drug: Mometasone nasal spray

INTERVENTIONS:
Drug: placebo
  Arms: placebo
Drug: Mometasone Nasal Spray
  Arms: NASONEX® Nasal Spray (Schering Corporation)
Drug: Mometasone nasal spray
  Arms: Mometasone Nasal Spray (Watson Laboratories, Inc)

SUMMARY:
A Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multi-Site Study to Compare the Clinical Equivalence of Mometasone Nasal Spray (Watson Laboratories, Inc) with NASONEX® Nasal Spray (Schering Corporation) in the Relief of the Signs and Symptoms of Seasonal Allergic Rhinitis

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant non-lactating female
* 12 years of age or older
* Signed informed consent form, which meets all criteria of current FDA regulations. For patients under the age of majority in the state the study is being conducted (18 years in most states) the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form that will be written in such a way as to be understandable to a child.
* If female and of child-bearing potential, have a negative urine pregnancy test and is prepared to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom with spermicide, IUD, oral, injected, transdermal or implanted hormonal contraceptives). In order for hormonal birth control to be considered a reliable method the patient must have been on their regimen for at least 28 days.
* Documented positive allergic skin test, performed within the previous 12 months, to one or more of the allergens in season at the time the study is being conducted.
* A minimum of two consecutive years of previous history of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* A score of at least 6 on the reflective Total Nasal Symptom Score (rTNSS) and a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms (see Appendix A) representing the 12 hours prior to the screening visit.
* An average composite score of at least 6 on the reflective Total Nasal Symptom Score (rTNSS) and a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms (see Appendix A) representing the last 3 days of the 7-day placebo run-in period before the randomization visit and the morning of the first day of the randomization visit.

Exclusion Criteria:

* Under 12 years of age.
* Females who are pregnant, lactating or likely to become pregnant during the study.
* Negative or lack of documented skin allergen test (performed within the previous 12 months) to at least one of the allergens in season at the time the study is being conducted. The results of all positive skin allergen test results should be reported.
* Patients who suffer from chronic signs and symptoms of Perennial Allergic Rhinitis (PAR) should be excluded from the study unless the Investigator assesses that the patient's current signs and symptoms are a clear exacerbation of Seasonal Allergic Rhinitis (SAR) rather than chronic PAR.
* Patients who suffer only from perennial allergic rhinitis or seasonal allergic rhinitis to a different allergen than that in season at the time the study is conducted.
* Previous history of less than 2 years of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* A total score of less than 6 on the reflective Total Nasal Symptom Score (rTNSS) or a score less than 2 for "nasal congestion" or a score less than 2 for all 3 of the remaining symptoms (see Appendix A). Any patient who meets the minimum rTNSS requirements at the start of the placebo lead-in period but no longer meets the requirements prior to the randomized active treatment period of the study cannot continue in the active treatment period.
* History of asthma over the previous two years that required chronic therapy. Occasional acute or mild exercise induced asthma will be allowable on the condition that the treatment of the attacks is restricted to beta-agonists only.
* Patients with nasal conditions, including infectious rhinitis, rhinitis medicamentosa or atrophic rhinitis.
* Clinically significant nasal deformity (e.g. significantly deformed septum, nasal polyps or ulcers) or any recent nasal surgery or trauma that has not completely healed.
* Sinus infection within the previous 30 days or history of re-occurring sinus infections.
* Patient has started immunotherapy (including topical or desensitization therapy) or changed their dose of immunotherapy within 30 days of the first placebo lead-in dose or is likely to have to start immunotherapy, or change their current dose during the study.
* Treatment for oral Candidiasis within 30 days of starting the study or a current oral Candidiasis infection.
* Upper respiratory tract infection within the previous 30 days.
* Patients with a history of tuberculosis.
* Patients with the presence of glaucoma, cataracts, ocular herpes simplex, conjunctivitis or other eye infection not related to the diagnosis of SAR within 14 days of enrollment.
* The patient has had recent exposure (30 days) or was at risk of being exposed to chicken pox or measles.
* Patients with any untreated fungal, bacterial, systemic viral infections within the previous 30 days.
* Use of any ophthalmic steroids within 14 days or nasal, inhaled or systemic steroids within 30 days of the study start. Super or high potency topical steroids should not be used during the study. The use of low potency topical corticosteroids (e.g. OTC 1% hydrocortisone) will be allowed. The use of hormonal contraceptives or hormone replacement therapy is allowed, on condition the patient has been on a stable dosing regimen for at least 28 days prior to the start of the study and remains on the same dosing regimen during the study.
* Use of intranasal or systemic second-generation anti-histamines (e.g. fexofenadine, loratadine, desloratadine, cetirizine) within 10 days of enrollment.
* Use of intranasal cromolyn within 14 days of enrollment.
* Use of intranasal or systemic first-generation anti-histamines, leukotriene receptor antagonists (montelukast) or other nasal decongestants within 3 days of enrollment.
* Use of any tricyclic anti-depressant within 30 days of enrollment.
* Patients with attention-deficit disorder being treated with methylphenidate containing products that have not been on a stable dosing regimen for at least the 30 previous days and who cannot remain on the same dosing regimen throughout the study.
* Desensitization therapy to the seasonal allergen that is causing the patients allergic rhinitis within the previous 6 months.
* Previous SAR and/or PAR that has proven unresponsive to steroid therapy.
* Any known hypersensitivity to mometasone, other steroids or any of the components of the study nasal spray.
* Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participating or could jeopardize the integrity of the study evaluations.
* Receipt of any drug as part of a research study within 30 days prior to the first placebo lead-in dose.
* Planned travel outside of the local area for more than 2 consecutive days or 3 days in total, during the patient's participation in the study.
* Previous participation in this study.
* The patient has a history of non-compliance with medication regimens or treatment protocols in previous clinical studies.
* The patient is a member of the investigational study staff or a member of the family of the investigational study staff.
* The patient currently smokes cigarettes, cigars, and/or pipes and is a heavy smoker (for example, on average more than 10 cigarettes per day).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Investigator site 18, Stockbridge, Georgia
  - Investigator site 1, Louisville, Kentucky
  - Investigator site 3, Bethesda, Maryland
  - Investigator Site 19, Minneapolis, Minnesota
  - Investigator Site 24, St Louis, Missouri
  - Investigator site 22, Bellevue, Nebraska
  - Investigator Site 23, Skillman, New Jersey
  - Investigator site 2, Corning, New York
  - Investigator site 9, High Point, North Carolina
  - Investigator site 20, Raleigh, North Carolina
  - Investigator site 25, Cincinnati, Ohio
  - Investigator site 21, Sylvania, Ohio
  - Investigator site 16, Spartanburg, South Carolina
  - Investigator Site 10, Austin, Texas
  - Investigator Site 12, Austin, Texas
  - Investigator site 6, Austin, Texas
  - Investigator Site 11, Kerrville, Texas
  - Investigator Site 7, New Braunfels, Texas
  - Investigator Site 13, San Antonio, Texas
  - Investigator site 14, San Antonio, Texas
  - Investigator site 5, San Antonio, Texas
  - Investigator site 8, San Antonio, Texas
  - Investigator site 4, Waco, Texas
  - Investigator Site 15, Draper, Utah
  - Investigator Site 17, Greenfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized subjects in active treatment.
Groups:
- Placebo: Placebo vehicle nasal spray (no active ingredients) Dose = 4 total actuations in alternating nostrils
- NASONEX® Nasal Spray (Schering Corporation); Mometasone Nasal Spray (Watson Laboratories, Inc): Mometasone Nasal spray, 50 mcg per actuation Dose = 4 total actuations in alternating nostrils (total dose = 200 mcg)
Period: Overall Study
Arm/Group | Placebo | NASONEX® Nasal Spray (Schering Corporation) | Mometasone Nasal Spray (Watson Laboratories, Inc)
Started | 175 | 350 | 355
Completed | 172 | 347 | 345
Not Completed | 3 | 3 | 10
Not completed — Early Visit Window | 0 | 1 | 4
Not completed — Enrolled in Error | 0 | 1 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Restricted Medication | 0 | 0 | 2
Not completed — Significant worstening of SAR | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NASONEX® Nasal Spray (Schering Corporation) | Mometasone Nasal Spray (Watson Laboratories, Inc) | Total
Number analyzed (Participants) | 175 | 350 | 355 | 880
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.31 (14.45) | 38.70 (14.45) | 38.80 (14.18) | 39.00 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 243 | 216 | 585
  Male | 49 | 107 | 139 | 295
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 123 | 259 | 276 | 658
  Black/African American | 45 | 75 | 68 | 188
  Asian | 5 | 11 | 9 | 25
  Native Hawaiian/Other Pacific Islander | 1 | 3 | 1 | 5
  Other | 1 | 2 | 1 | 4
Tobacco Use [Count of Participants; unit: Participants]
  Have used tobacco | 7 | 14 | 13 | 34
  Have not use tobacco | 168 | 336 | 342 | 846
Primary Allergen [Count of Participants; unit: Participants]
  Tree | 110 | 234 | 231 | 575
  Multi-Allergen | 64 | 114 | 119 | 297
  Grass | 1 | 2 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average AM/PM Reflective Total Nasal Symptom Score (rTNSS) Over Days 1 to 14.
Description: The Total Nasal Symptom Score Scale was used. Patients rated each of the following four symptoms on a scale from 0 to 3 : Nasal Congestion, Runny Nose, Sneezing, and Itchy Nose. Measurements were taken twice daily approximately 12 hours apart.
  0= No symptom
  1. Mild symptoms (sign/symptom present, minimal awareness, easily tolerated)
  2. Moderate symptom (definite awareness of sign/symptom, bothersome but tolerable)
  3. Severe symptom (sign/symptom hard to tolerate, causes interference with daily activities and/or sleeping)
Time Frame: Twice daily from Baseline to 2 weeks
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- NASONEX® Nasal Spray (Schering Corporation): Mometasone Nasal spray, 50 mcg per acuation Dose = 4 total actuations in alternating nostrils (total dose = 200 mcg)
Arm/Group | NASONEX® Nasal Spray (Schering Corporation) | Mometasone Nasal Spray (Watson Laboratories, Inc)
Number analyzed (Participants) | 346 | 342
score on a scale | 1.861 (2.186) | 1.600 (2.223)
Statistical Analysis 1: Comparison: NASONEX® Nasal Spray (Schering Corporation) vs Mometasone Nasal Spray (Watson Laboratories, Inc); Conducted on Per Protocol Population; Test type: Equivalence — Equivalence based on Test/Reference Ratio and 90% confidence interval (as per OGD guidance); Ratio Test/Reference LS Mean = 114.723, 90% CI 2-sided [99.077 to 134.286]

2. Primary Outcome: Superiority of Active Treatment Arms Over Placebo
Description: Superiority analysis of Change From Baseline in rTNSS for both active arms compared to placebo arm. The Total Nasal Symptom Score Scale was used. Patients rated each of the following four symptoms on a scale from 0 to 3: Nasal Congestion, Runny Nose, Sneezing, and Itchy Nose twice daily approximately 12 hours apart.
  0= No symptom
  1. Mild symptoms (sign/symptom present, minimal awareness, easily tolerated)
  2. Moderate symptom (definite awareness of sign/symptom, bothersome but tolerable)
  3. Severe symptom (sign/symptom hard to tolerate, causes interference with daily activities and/or sleeping)
Time Frame: Twice daily from Baseline to 2 weeks
Population: Intent to treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | NASONEX® Nasal Spray (Schering Corporation) | Mometasone Nasal Spray (Watson Laboratories, Inc)
Number analyzed (Participants) | 173 | 348 | 354
score on a scale | 0.898 (1.762) | 1.609 (2.225) | 1.863 (2.191)
Statistical Analysis 1: Comparison: Placebo vs Mometasone Nasal Spray (Watson Laboratories, Inc); The superiority of treatment over the placebo will be concluded if the treatment's mean change from baseline is statistically significantly greater (p<0.05, 2-sided) than that of the placebo in the ANCOVA based on the treatment and placebo results. The superiority of Test and Reference treatments over the placebo will be evaluated identically in a separate ANCOVA; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs NASONEX® Nasal Spray (Schering Corporation); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0002, ANCOVA

ADVERSE EVENTS:
Time Frame: AEs were collected from ICF signature until end of study (~1 month in duration).
Arm/Group | Placebo | NASONEX® Nasal Spray (Schering Corporation) | Mometasone Nasal Spray (Watson Laboratories, Inc)
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/350 | 0/355
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/350 | 0/355
Other Adverse Events (participants affected / at risk) | 20/175 | 23/350 | 18/355
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=175) | NASONEX® Nasal Spray (Schering Corporation) (N=350) | Mometasone Nasal Spray (Watson Laboratories, Inc) (N=355)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1)
Hyperthryroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular Hyperaemia (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes Simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Sinus Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other